CLINICAL TRIAL: NCT03717298
Title: Evaluation of the Effect of Ocoxin-Viusid® Nutritional Supplement in the Life Quality in Patients Diagnosed With Advanced Pancreatic Adenocarcinoma. Phase II
Brief Title: Evaluation of Ocoxin-Viusid® in Advanced Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OOS-CANCER-6
Record Dates: First submitted 2018-09-28; First posted 2018-10-24 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Adenocarcinoma of the Pancreas; Pancreatic Cancer; Advanced Cancer; Digestive System Neoplasms; Pancreatic Neoplasms; Endocrine Gland Neoplasms; Digestive System Diseases; Endocrine System Diseases; Pancreatic Diseases
Keywords: Nutritional supplement; Advanced Pancreatic adenocarcinoma; Ocoxin-Viusid; Oxidative stress; Antioxidant
MeSH Terms: conditions — Pancreatic Neoplasms; Digestive System Neoplasms; Endocrine Gland Neoplasms; Digestive System Diseases; Endocrine System Diseases; Pancreatic Diseases | interventions — Ocoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ocoxin-Viusid (Experimental): It will be used at a rate of 60 ml daily (1 vial every 12 hours).
  Interventions: Dietary Supplement: Ocoxin-Viusid®

INTERVENTIONS:
Dietary Supplement: Ocoxin-Viusid® — An oral solution of Ocoxin-Viusid® (30 ml vials) will be used at a rate of 60 ml daily (1 vial every 12 hours), preferably administered after breakfast and lunch. It will be prescribed for a period of 2 weeks before starting the QT.
  The treatment with Ocoxin-Viusid® will continue in the possible periods of time of suspension of the chemotherapy treatment due to toxicities attributable to the oncospecific treatment.
  The treatment will be administered continuously from the inclusion of the patient in the study, up to one year.

SUMMARY:
The investigators hypothesized that with the administration of the nutritional supplement Ocoxin-Viusid® is expected to improve the quality of life and enhance tolerance to chemotherapy in at least 70% of patients diagnosed with advanced pancreatic adenocarcinoma, treated at the "Hermanos Ameijeiras" Surgical Clinical Hospital. Phase II clinical trial, open, multicenter, nonrandomized.

DETAILED DESCRIPTION:
To assess the effect of Ocoxin-Viusid® on the quality of life of patients with advanced pancreatic adenocarcinoma.

To evaluate the effect of Ocoxin-Viusid® on the quality of life of patients. To evaluate the influence of Ocoxin-Viusid® on tolerance to onco-specific therapy.

Identify the changes that occur in the nutritional status of patients receiving the supplement.

To evaluate the toxicity of Ocoxin-Viusid® in combination with chemotherapy in patients with advanced pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any sex, resident in Cuba, with an age greater than or equal to 18 years.
* Patients that meet the diagnostic criteria.
* Patients with general health according to Karnofsky ≥70 %.
* Life expectancy greater than or equal to 3 months.
* Patients eligible to receive chemotherapy.
* Patients who have signed the informed consent.
* Patients who have laboratory values in parameters that do not contraindicate the administration of chemotherapy:
* Hemoglobin ≥ 90 g / l.
* Total Leukocyte Count ≥ 3.0 x 109 / L.
* Absolute Neutrophil Count ≥1.5 x 109 / L.
* Platelet count ≥100 x 109 / L.
* Total bilirubin values ≤ 1.5 times the upper limit of the normal range established in the institution.
* TGO and TGP values ≤2.5 times the upper limit of the normal interval established in the institution.
* Creatinine values within the normal limits of the institution.

Exclusion Criteria:

* Pregnant or lactating patients.
* Patients with known hypersensitivity to any of the active ingredients of the chemotherapy used
* Patients who are receiving another product under investigation.
* Patients with decompensated intercurrent diseases, including: hypertension, diabetes mellitus, ischemic heart disease, active infections, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, liver damage or any other special condition that at the discretion of the doctor puts their health at risk and his life during the study or his participation in the trial.
* Patients with brain metastases.
* Patients with mental disorders that may limit adherence to the requirements of the clinical trial and may hinder the collection of information, treatment or follow-up.

It is planned to include a total of 30 patients in the study, taking into account 10% of losses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Quality of Life: EORTC QLQ-C30 | 12 months
  Life quality measurement through the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 30 (ORTC QLQ-C30): an integrated system for assessing the healthrelated quality of life (QoL) of cancer patients participating in international clinical trials. It's composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.

SECONDARY OUTCOMES:
Nutritional Status of the patient during Chemotherapy | 12 months
  Variations in the patient's nutritional status will be considered, measured by body mass Index (a measure of body fat based on height and weight that applies to adult men and women)
Adverse Events-AE during Chemotherapy Test | 12 months
  A test with the following questions:
  Occurrence of an AE in the subject [Yes, No]; Description of the AE [Name of the event]; Duration of the AE [Difference between the start and end date of the event]; Intensity of the AE [According to CTCAE version 4 it will classify in Light, Moderate, Severe, Life-threatening consequences, Death related to AE]; Seriousness of the AE [serious or not serious], Attitude with respect to the treatment under study [No changes, dose modification, temporary or definitive interruption of the study treatment], Result of the AE [recovered, improved, persisted or sequelae], Causal relationship [According to WHO algorithm it will classify in very probable, probable, possible, improbable, unrelated, not evaluable]
Hematology test | 12 months
  Levels of Hemoglobin, Platelets, Hemogram with differential in blood extractions.
Blood Chemistry test | 12 months
  Measure levels of GPT, GOT, Creatinine, Glycemia, Bilirrubin, Alkaline Phosphatase, LDH in blood.
Compliance with the treatment with chemotherapy (CT) and Immunotherapy (IT) test | 12 months
  Test with the next parameters: if the administration of chemotherapy (CT) and Immunotherapy (IT) treatments will be considered at planned time, number of the cycle administered out of date, days elapsed since the previous cycle and, cause that caused the administration of the CT/IT outside the planned date. In the case of the dose, the medication in which it was modified will be taken into account, as well as the modified dose.

CONTACTS AND LOCATIONS:
Locations (1):
- "Hermanos Ameijeiras" Surgical Clinical Hospital, La Habana, Cuba

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Burris HA 3rd, Moore MJ, Andersen J, Green MR, Rothenberg ML, Modiano MR, Cripps MC, Portenoy RK, Storniolo AM, Tarassoff P, Nelson R, Dorr FA, Stephens CD, Von Hoff DD. Improvements in survival and clinical benefit with gemcitabine as first-line therapy for patients with advanced pancreas cancer: a randomized trial. J Clin Oncol. 1997 Jun;15(6):2403-13. doi: 10.1200/JCO.1997.15.6.2403. PMID 9196156
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Tobita K, Kijima H, Dowaki S, Kashiwagi H, Ohtani Y, Oida Y, Yamazaki H, Nakamura M, Ueyama Y, Tanaka M, Inokuchi S, Makuuchi H. Epidermal growth factor receptor expression in human pancreatic cancer: Significance for liver metastasis. Int J Mol Med. 2003 Mar;11(3):305-9. PMID 12579331
- [Background] Burris H 3rd, Rocha-Lima C. New therapeutic directions for advanced pancreatic cancer: targeting the epidermal growth factor and vascular endothelial growth factor pathways. Oncologist. 2008 Mar;13(3):289-98. doi: 10.1634/theoncologist.2007-0134. PMID 18378539
- [Background] Ueda S, Ogata S, Tsuda H, Kawarabayashi N, Kimura M, Sugiura Y, Tamai S, Matsubara O, Hatsuse K, Mochizuki H. The correlation between cytoplasmic overexpression of epidermal growth factor receptor and tumor aggressiveness: poor prognosis in patients with pancreatic ductal adenocarcinoma. Pancreas. 2004 Jul;29(1):e1-8. doi: 10.1097/00006676-200407000-00061. PMID 15211117
- [Background] Korc M, Meltzer P, Trent J. Enhanced expression of epidermal growth factor receptor correlates with alterations of chromosome 7 in human pancreatic cancer. Proc Natl Acad Sci U S A. 1986 Jul;83(14):5141-4. doi: 10.1073/pnas.83.14.5141. PMID 3014534
- [Background] Immervoll H, Hoem D, Kugarajh K, Steine SJ, Molven A. Molecular analysis of the EGFR-RAS-RAF pathway in pancreatic ductal adenocarcinomas: lack of mutations in the BRAF and EGFR genes. Virchows Arch. 2006 Jun;448(6):788-96. doi: 10.1007/s00428-006-0191-8. Epub 2006 Apr 6. PMID 16598499
- [Background] Lee J, Jang KT, Ki CS, Lim T, Park YS, Lim HY, Choi DW, Kang WK, Park K, Park JO. Impact of epidermal growth factor receptor (EGFR) kinase mutations, EGFR gene amplifications, and KRAS mutations on survival of pancreatic adenocarcinoma. Cancer. 2007 Apr 15;109(8):1561-9. doi: 10.1002/cncr.22559. PMID 17354229
- [Background] Russo A, Rizzo S, Bronte G, Silvestris N, Colucci G, Gebbia N, Bazan V, Fulfaro F. The long and winding road to useful predictive factors for anti-EGFR therapy in metastatic colorectal carcinoma: the KRAS/BRAF pathway. Oncology. 2009;77 Suppl 1:57-68. doi: 10.1159/000258497. Epub 2010 Feb 2. PMID 20130433
- [Background] da Cunha Santos G, Dhani N, Tu D, Chin K, Ludkovski O, Kamel-Reid S, Squire J, Parulekar W, Moore MJ, Tsao MS. Molecular predictors of outcome in a phase 3 study of gemcitabine and erlotinib therapy in patients with advanced pancreatic cancer: National Cancer Institute of Canada Clinical Trials Group Study PA.3. Cancer. 2010 Dec 15;116(24):5599-607. doi: 10.1002/cncr.25393. Epub 2010 Sep 7. PMID 20824720